CLINICAL TRIAL: NCT03761485
Title: Dental Fluorosis Risk by the Use of Acidulated Fluoride Dentifrice: Clinical Trial - Epidemiological Study With Children Residing in an área Without Public Water Fluoridation
Brief Title: Dental Fluorosis Risk by the Use of Acidulated Fluoride Dentifrice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Fabio Correia Sampaio, Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Acidulated fluoride dentifrice
Record Dates: First submitted 2018-08-25; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Caries, Dental; Fluorosis, Dental
MeSH Terms: conditions — Dental Caries; Fluorosis, Dental

STUDY DESIGN:
Intervention Model Description: Randomized double blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dentifrice 750 ppm of NaF acidulated (Experimental): Use of Dentifrice Fluoride Use of few of dentifrice on brushing for 12 months
  Interventions: Other: Use of Dentifrice Fluoride
- Dentifrice 1.100 ppm of NaF neutral (Active Comparator): Use of Dentifrice Fluoride Use of few of dentifrice on brushing for 12 months
  Interventions: Other: Use of Dentifrice Fluoride
- Dentifrice 1.100 ppm of NaF acidulated (Active Comparator): Use of Dentifrice Fluoride Use of few of dentifrice on brushing for 12 months
  Interventions: Other: Use of Dentifrice Fluoride

INTERVENTIONS:
Other: Use of Dentifrice Fluoride — Use of few of dentifrice on brushing during a year

SUMMARY:
This research aimed to evaluate the risk of dental fluorosis by using an experimental fluoridated acidulated dentifrice compared to conventional dentifrices in two-to-four-year-old children residing in a non fluoridated area by the concentration of fluoride incorporated in childrens' nails, as well as the incorporation of F into the biofilm. Two hundred and ten children participated on this study. They were randomly allocated into three groups differing according to the type of dentifrice used over 12 months: G1:1100 ppm F, pH 4.5; G2:750 ppm F, pH 4.5; G3:1100 ppm F, pH 7.0. The dentifrice was placed on the toothbrush using the "drop" technique. The toenails of the biggest toe were collected in three moments, corresponding to the experimental period of use of the dentifrices (T1, T2 and T3), as well as the biofilm which was collected twice, 5 and 60 minutes after brushing. The nails and biofilm fluoride concentration were analyzed on a specific electrode using the HMDS diffusion facilitated technique.

DETAILED DESCRIPTION:
This is a randomized, double-blind, interventional trial, adopting a strategy for collecting data, collecting data from the children's biofilm. This study was carried out in three Child Education Reference Centers (CREIs) located in different points of the city of João Pessoa PB.

The city is located in the Northeast region of Brazil, on the coast of the state of Paraíba and has about 600 thousand inhabitants (IBGE, 2013). João Pessoa has already had fluoridated water for a period of two years until the mid-1980s, but so far the project has been deactivated.

The 452 children participating in the study were divided into three groups according to the dentifrice used in a 12 - month period: G1: 1,100 ppm F - pH 4.5; G2: 750 ppm F-pH 4.5; and G3: 1100 ppm F-pH 7.0. The toothpaste was supplied by Oralls (São Jose dos Campos-SP, Brazil) and dental brushes by Bitufo (Hypermarcas, São Paulo, SP-, Brazil) and there was no conflict of interest. For the random distribution of the groups, the CREIs were considered as units, so that only one type of toothpaste was distributed in each CREI, thus facilitating the control of the dentifrices delivery by the teachers, as well as the supervised brushing in CREI itself.

The toenails of the biggest toe were collected in three moments, corresponding to the experimental period of use of the dentifrices (T1, T2 and T3), as well as the biofilm which was collected twice, 5 and 60 minutes after brushing. The nails and biofilm fluoride concentration were analyzed on a specific electrode using the HMDS diffusion facilitated technique.

Nails of the large toes were collected because they provide a sufficient nail mass for analysis and because there has been a reported possibility of contamination of the toenails (Buzalaf, Pessan et al., 2006). The nail samples of each child were cleaned with deionized water using a dental brush, taken to the ultrasound apparatus with deionized water for 10 min, dried at 60 ± 5 ° C and weighed on the analytical balance The presence of F was analyzed as described in the previous item, according to the method of Taves (1968), as modified by Whitford (1996). F patterns (0.00475, 0.0095, 0.019, 0.095, 0.190 and 0.95 mg F) were prepared by serial dilution of a stock solution of 0.1 MF (Orion) in triplicate and diffused in the same manner as the samples. The average repeatability of the readings based on duplicate samples was 95%. Whenever the sample weight was> 20 mg, the analysis was performed in duplicate.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 2 to 4 years of age of both sexes
* Who were enrolled in one of the 3 CREIs that participated in the research
* Presence of deciduos teeth

Exclusion Criteria:

* Presented high mobility of the children (incompatible with the planning of a longitudinal study)
* Children who did not allow the clinical examination in the school
* Children using orthodontic appliances or children with extensive caries lesions with dentin sensitivity
* Children not residing in the city of João Pessoa-PB from birth to 4 years due to the fluoridation of water from public supply.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 452 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Concentration of intraoral fluoride | 1 year
  Effective of capacity to concentration of fluoride in biofilm (ppm)
Effect of intraoral fluoride - software | 1 year
  Reduction of initial lesions carie give by mm² analysed by software
Effect of intraoral fluoride | 1 year
  Reduction of initial lesions carie give by visual scale (Nyvad scale)
Concentration of nail fluorid | 1 year
  Concentration of fluoride in nail (ppm)

IPD SHARING:
Plan to Share IPD: No